CLINICAL TRIAL: NCT01318330
Title: Five-Week, Multi-center, Phase I Clinical Trial to Evaluate Safety of Homeo-GH After Intra Venus Administration for the Treatment of Graft Versus Host Disease Patients
Brief Title: Safety Study of Homeo-GH (Bone Marrow Derived Clonal Mesenchymal Stem Cell) to Treat Acute/Chronic Graft Versus Host Disease (GVHD)
Acronym: Homeo-GH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HomeoTherapy Co., Ltd (Industry)
Responsible Party: Sun U. Song/Ph.D/Professor, Inha Univ. College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Homeo-GH
Record Dates: First submitted 2011-03-14; First posted 2011-03-18 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2011-03

CONDITIONS: Graft-vs-Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Homeo-GH — Bone Marraw derived Clonal Mesenchymal Stem Cell (cMSC)

SUMMARY:
Official Title: Five-Week, Multi-center, Phase I Clinical Trial to Evaluate Safety of Homeo-GH after Intra Venus Administration for the Treatment of Graft versus Host Disease Patients

Sponsor: HomeoTherapy Co.,Ltd

Study Design: Single Group, Open Label, 5 Week, Safety Study

This study is designed to evaluate the safety of ex-vivo cultured adult human clonal mesenchymal stem cells (cMSC) derived from human bone marrow in subjects experiencing acute or chronic graft-versus-host disease (GVHD).

Study Type: Interventional

DETAILED DESCRIPTION:
Allogeneic MSCs being used in current human clinical trials are nonclonal, i.e., such MSCs may have other types of cells in the final stem cell product. Some concerns exist about the heterogeneity of these nonclonal MSCs that are isolated and expanded by the conventional density-gradient centrifugation method. Recently, we developed a new protocol, called the subfractionation culturing method (SCM), to generate single-cell-derived clonal MSC (cMSC) lines from whole bone marrow aspirate without employing any centrifugation step for mononuclear cells and enzyme treatment process. This method allowed us to rapidly establish single-cell-derived human clonal MSC (hcMSC) lines from raw bone marrow aspirates and to establish a library of these hcMSC lines (Song et al., 2008).

The goal of this study is to evaluate the safety of allogeneic cMSCs established by the SCM and manufactured in GMP facility. This phase I clinical trial is a multicenter, single dose study of cMSC (1 x 10e6 cMSCs/Kg recipient's bodyweight). Clonal MSCs will be infused to acute or chronic GVHD patients via an intravenous injection. Every patients will receive the same treatment

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from patient
* Patients with ages greater than 18 years
* Neutrophill count > 1,000 cells/mm3
* Adequated cardiac function with no evidence of cardiac disease
* Patients who had complete remission after bone marrow transplantation
* Patients who can sign an informed consent form by him- or her-self or legal representative

Exclusion Criteria:

* Patients with unstable transplant after bone marrow transplantation
* Patients with unstable vital sign
* Patients with positive penicillin skin test
* Patients who had transplantation to treat solid tumor
* Patients with bacterial, viral or fungal infection not being controlled by the adequate treatment (more than moderate infection)
* Patients who, in the investigator's point of view, are not in proper state for the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate number of paticipants with adverse events | Within the first 5 week
  Aderse Events were record relationship with Investigational Product
  * Not related
  * Unlikely
  * Possible
  * Probable
  * High probable
  The severity of adverse events were graded refer to CTCAE (Common Terminology Criteria for Adverse Events) Ver.4.0

SECONDARY OUTCOMES:
GVHD clinical response | Within the first 5 week
  Clinical response was evaluated base on GVHD grding system
  * CR (Complete Response)
  * PR (Partial Response)
  * SD (Stable Disease)
  * PD (Progressive Disease)

CONTACTS AND LOCATIONS:
Overall Officials: SunUk Song, Ph.D., Study Director — Inha Univ. College of Medicine; Charles, JH Kim, Ph.D., Study Director — HomeoTherapy Co., Ltd; Hyun Gyu Lee, M.D.,Ph.D., Principal Investigator — Inha Univerisity Hospital
Locations (4):
- South Korea (4):
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul